CLINICAL TRIAL: NCT06625385
Title: A Post-market, Prospective, Multi-center, Single-arm Study Evaluating the Safety and Efficacy of the 3M™ V.A.C. Peel and Place Dressing Used in Conjunction With 3M™ V.A.C.® Therapy
Brief Title: A Study Evaluating the Safety and Efficacy of the 3M™ V.A.C. Peel and Place Dressing
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Solventum US LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EM-05-015140
Record Dates: First submitted 2024-09-12; First posted 2024-10-03 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Wound
Keywords: Open; Closed
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- 3M™ V.A.C.® Peel and Place Dressing (Experimental): 3M™ V.A.C.® Peel and Place Dressing used in conjunction with 3M™ V.A.C.® Therapy
  Interventions: Device: 3M™ V.A.C.® Peel and Place Dressing

INTERVENTIONS:
Device: 3M™ V.A.C.® Peel and Place Dressing — Application of 3M™ V.A.C.® Peel and Place Dressing used in conjunction with 3M™ V.A.C.® Therapy

SUMMARY:
The purpose of this clinical study is to obtain post-market safety and efficacy data when the V.A.C.® Peel and Place dressing is used in conjunction with 3M™ V.A.C.® Therapy.

DETAILED DESCRIPTION:
This is a prospective, post-market, multi-center, single-arm study. A target of 90 enrolled Subjects with 1 enrolled study wound per Subject is planned for this study, including 60 open wounds (10 for each type of open wound) and 30 closed or covered wounds (10 for each type of closed/covered wound). The entire duration of the study is expected to last approximately 2 years. Individual Subject participation is expected to last up to 20 days, including a screening period lasting up to 5 days, the day of initial treatment, dressing change visits as clinically appropriate but no more than 7 days from dressing application, and an end-of-treatment (EOT)/end-of-study (EOS) visit between Day 7 and Day 14 after the initial dressing application.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is at least 22 years old at the time of consent.
2. Subject or legally authorized representative (LAR) is able to provide informed consent.
3. Subject has a wound deemed appropriate for treatment with a V.A.C.® Peel and Place dressing (used in conjunction with 3M™ V.A.C.® Therapy), according to the instructions for use for the dressing, including the following wound types:

   * an open wound: acute/traumatic wound, dehisced surgical wound within 30 days of surgery, burn, venous ulcer, diabetic ulcer, or pressure ulcer Note: Prior to initial placement, the wound may be debrided, as clinically indicated
   * a closed or covered wound secured with sutures or staples: closed surgical incision, skin flap closure, or skin graft (recipient site)
4. Subject is willing and able to attend all study visits.

Exclusion Criteria:

1. Subject is pregnant or lactating prior to application of the initial dressing. *

   *Women who have had surgical sterilization by a medically accepted method (ie, tubal ligation, hysterectomy, or oophorectomy) or are post-menopausal, defined as not having menstruation for > 12 months will not be required to undergo pregnancy testing.
2. Subject is participating in another interventional clinical study or was enrolled in a clinical trial within the last 30 days before screening.
3. Subject has been diagnosed with a malignancy in the wound.
4. Subject has untreated osteomyelitis or untreated cellulitis in the wound.
5. Subject has an untreated systemic infection.
6. Subject has active cellulitis in the peri-wound area.
7. Subject has a known allergy or hypersensitivity to study materials: dressing(s), and/or dressing components such as acrylic or silicone adhesives or polyurethane.
8. Subject has, in the opinion of the investigator, a clinically significant condition that would impair the Subject's ability to comply with the study procedures or would compromise assessment of endpoints (wound/peri-wound condition).
9. Subject has had radiation directly to the wound area.
10. Subject received hyperbaric oxygen therapy within 30 days before the initial application of a V.A.C.® Peel and Place dressing.
11. Subject has been diagnosed with a major vascular deficit limiting arterial inflow into the wound region, as determined by the investigator's interpretation of the subject's medical history.
12. In the case of a lower extremity wound, the Subject has one of the following:

    * an ankle brachial index < 0.8;
    * no palpable pulse; or
    * no discernable audio Doppler signal. Individual wounds are to be excluded from the study if they meet any of the following criteria

1. Wound has necrotic tissue and/or eschar present. NOTE: After debridement of necrotic tissue and complete removal of eschar, the V.A.C.® Peel and Place dressings may be used.

2. Wound contains a non-enteric or unexplored fistula(s) in the wound bed. 3. Wound has tunneling. 4. Wound has undermining that is ≥ 2 cm in any direction from the wound edge. 5. Wound site has inadequate hemostasis, as determined by the investigator. 6. Wound has exposed vessels, anastomotic sites, organs, or nerves that cannot be protected prior to placement of the V.A.C.® Peel and Place Dressings.

7. Wound has a depth greater than 2 cm (for small dressings), 4 cm (for medium dressing size), or 6 cm (for the large dressing size).

8. The wound received, within 30 days before initiating V.A.C.® Therapy, treatment with any of the following:

* any previous negative pressure wound therapy device.
* growth factors.
* bioengineered tissue products, eg, skin or dermal substitutes. 9. Wound was closed with tissue adhesive. 10. Wound has, in the opinion of the Investigator, any characteristic that would make it unsuitable for the study.

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-01-20 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of (ADEs) | 14 days
  The incidence of adverse device effects (ADEs)

SECONDARY OUTCOMES:
Percentage of closed surgical incisions and skin flaps that remain closed | 14 days
  The percentage of closed surgical incisions and skin flaps that remain closed throughout treatment
Percentage of skin grafts with ≥ 90% graft take | 14 days
  The percentage of skin grafts with ≥ 90% graft take at the end of treatment
Percentage of open wounds with evidence of healing | 14 days
  The percentage of open wounds with evidence of healing, as evidenced by any of the following:
  * decrease in total wound area (cm2) from baseline to the end of treatment,
  * decrease in total wound volume (cm3) from baseline to the end of treatment,
  * decrease in average wound depth from baseline to the end of treatment,
  * increase in the percentage of the wound with red color composition (signifying healthy, viable tissue), from baseline to the end of treatment,
  * improved score for exudate amount from the first dressing change to the end of treatment
  * improved score for peripheral tissue edema from baseline to the end of treatment
  * new epithelialization from baseline to the end of treatment, or
  * wound is deemed ready for closure (via delayed primary closure, graft, or flap) at any time from baseline to the end of treatment
Overall rate of wound healing for both open wounds and closed/covered wounds | 14 days
  The overall rate of wound healing for both open wounds and closed/covered wounds, as evidenced by the aforementioned criteria

OTHER OUTCOMES:
Pain score associated with dressing removal | 14 days
  The pain score associated with dressing removal (ie, during dressing changes and at final dressing removal) - Subject-reported and based on the highest level of perceived pain.
  Whereby a score of 0 is indicative of "no pain" and a score of 10 indicates the "worst pain possible".

CONTACTS AND LOCATIONS:
Overall Officials: Sher-ree Beekman, Study Director — Solventum
Locations (3):
- United States (3):
  - IU Health Methodist Hospital, Indianapolis, Indiana
  - Washington University - Barnes Jewish Hospital, St Louis, Missouri
  - St. Luke's University Hospital, Bethlehem, Pennsylvania

IPD SHARING:
Plan to Share IPD: No